CLINICAL TRIAL: NCT02488421
Title: Real Evidence of Anticoagulation Treatment in Non-valvular Atrial Fibrillation in Germany, UK and France: REACT-AF 2
Brief Title: Real Evidence of Anticoagulation Treatment in Non-valvular Atrial Fibrillation in Germany, UK and France: REACT-AF2
Acronym: REACT-AF2
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: IMS Health (Other); OXON Epidemiology (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-371
Record Dates: First submitted 2015-06-18; First posted 2015-07-02 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Non-valvular Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Patient treated with Apixaban
- Patient treated with Rivaroxaban
- Patient treated with Dabigatran
- Patient treated with vitamin K antagonists

SUMMARY:
The purpose of this study is to determine and compare the persistence rate of newly prescribed apixaban, rivaroxaban, dabigatran and VKAs in patients with NVAF.

DETAILED DESCRIPTION:
Actual number of patients enrolled for UK : 15242 patients

Actual number of patients enrolled for Germany : 22880 patients

ELIGIBILITY:
Inclusion Criteria:

* Have an apixaban, rivaroxaban, dabigatran or VKA prescription during the study period
* Are ≥18 years old at index date
* Have ≥12 months of computerised medical data prior to index date
* Have a record of AF on or ever prior to index date (index OAC prescription)

Exclusion Criteria:

* Have a record for a valvular condition (ie, rheumatic valvular disease and prosthetic valves) on or ever prior to index date
* Have a history (ever prior to index date) of the Oral anticoagulant (OACs) which are prescribed during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 38122 (Actual)
Dates: Start 2014-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Persistence rate of newly prescribed apixaban, rivaroxaban, dabigatran and vitamin K antagonists (VKAs) in patients with non-valvular atrial fibrillation(NVAF) | 23 months for the UK and Germany, 25 months for France
  We defined non-persistence in the databases as the absence of index prescription for twice the median prescription duration; and calculated cumulative incidence (95% CIs) of persistence at the end of follow-up and at different time points after treatment initiation (3, 6, and 12 months)

SECONDARY OUTCOMES:
Demographic characteristics (Age, Gender, Smoking status, region of practice, data source) of patients with newly prescribed oral anticoagulants | 23 months for the UK and Germany, 25 months for France
Clinical characteristics (History of bleeding, myocardial infarction, stroke, Thromboembolism, congestive heart failure, vascular disease, hypertension, CHA2DS2-VASc score, HAS-BLED score, etc) of patients with newly prescribed oral anticoagulants | 23 months for the UK and Germany, 25 months for France
Adherence to newly prescribed oral anticoagulants based on Medication possession ratio (MPR) | 23 months for the UK and Germany
Compare persistence rates across oral anticoagulant therapies | 23 months for the UK and Germany, 25 months for France

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- [Derived] Collings SL, Vannier-Moreau V, Johnson ME, Stynes G, Lefevre C, Maguire A, Asmar J, Bizouard G, Duhot D, Mouquet F, Fauchier L. Initiation and continuation of oral anticoagulant prescriptions for stroke prevention in non-valvular atrial fibrillation: A cohort study in primary care in France. Arch Cardiovasc Dis. 2018 May;111(5):370-379. doi: 10.1016/j.acvd.2017.10.003. Epub 2018 Feb 3. PMID 29398546
- [Derived] Johnson ME, Lefevre C, Collings SL, Evans D, Kloss S, Ridha E, Maguire A. Early real-world evidence of persistence on oral anticoagulants for stroke prevention in non-valvular atrial fibrillation: a cohort study in UK primary care. BMJ Open. 2016 Sep 26;6(9):e011471. doi: 10.1136/bmjopen-2016-011471. PMID 27678530
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx